CLINICAL TRIAL: NCT05838027
Title: Philly Family Trust Study: A Pilot Randomized Controlled Trial of an Unconditional Cash Transfer to Improve Health Behaviors Among Adults With Chronic Diseases
Brief Title: Pilot Guaranteed Income Study, Philadelphia, April 2023
Acronym: PGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 852028; 5P30AG034546-14 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: At the end of the baseline assessment, participants will be randomized using a permuted block technique with block size of 4 to either usual care (Arm 1) or to the unconditional cash transfer intervention (Arm 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention
- Cash Transfer (Experimental): Participants will receive $125 every 2 weeks for 8 payments via ClinCard, for a total of $1000.
  Interventions: Behavioral: Cash Transfer

INTERVENTIONS:
Behavioral: Cash Transfer — Participants will receive $125 every 2 weeks for 8 payments via ClinCard, for a total of $1000.
  Arms: Cash Transfer

SUMMARY:
The goal of this pilot clinical trial is to learn about the effects of a short-term unconditional cash transfer (UCT) in people living with poverty and chronic disease (either prediabetes/diabetes or hypertension). The main questions it aims to answer are:

* How feasible and acceptable is the intervention?
* How are key health behaviors and outcomes affected by the intervention?
* What are reasonable effect sizes to expect in a larger trial?

Participants will complete surveys and health measurements at two timepoints 3 months apart. Half of the participants will be randomly assigned to the treatment where they will receive a UCT of $1000 over 4 months. Researchers will compare the treatment group to the control group to see if there are improvements in health risk factors directly related to insufficient resources (food and utility security, stress-levels, mental bandwidth), financial outcomes, and health behaviors.

DETAILED DESCRIPTION:
Health behaviors are major, modifiable risk factors for the development and progression of chronic diseases, which account for a large proportion of all deaths in the US and contribute to disparities in premature mortality based on both income and race. There is substantial evidence, for example, that behaviors like smoking, physical inactivity, and unhealthy diet are associated with an increased risk of cardiovascular disease (CVD), as are modifiable factors such as blood pressure, cholesterol, body mass index, and fasting glucose. A growing body of research suggests that poverty may affect health behaviors through financial and psychological pathways. However, few studies have rigorously examined the effects of poverty alleviation interventions on health behaviors, particularly among individuals at high risk for CVD. Even fewer studies have examined potential psychological mechanisms by which anti-poverty interventions might influence health behavior. This pilot project will examine the effect of unconditional cash transfers, an economic intervention that is gaining traction among policymakers, on risk factors for CVD and other chronic diseases. The project will focus on low-income adults in Philadelphia who have at least one health risk factor for CVD (diabetes/pre-diabetes and/or hypertension) and examines whether short-term, unconditional cash transfer payments result in changes in objective and self-reported health outcomes. The second aim examines potential psychological mechanisms through which the cash transfer intervention may affect study participants' behavior, including mental health, psychosocial stress, bandwidth, and future orientation. The third aim uses qualitative methods to understand participants' experiences with this study. The project activities will include developing and testing the cash transfer intervention (Stage 1) as well as basic science analysis of mechanisms of change (Stage 0).

Survey and measurement data will be collected from 100 participants at baseline and 3 month follow-up in a two-arm randomized controlled trial (50 in control, 50 in intervention). 16 participants will receive a blood pressure cuff to take home and send measurements weekly to assess the feasibility of at-home measurement (8 control, 8 intervention; half of each group will transmit wirelessly, the other half will not). 30 participants from the 3-month follow-up who are interested in doing an interview will provide additional qualitative data on their experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Pennsylvania Medicaid enrollee
* At least one recent clinic visit at Penn Family Care (earliest six months before start of recruitment)
* Diagnosis of pre-diabetes/diabetes and/or hypertension
* Actively prescribed a medication for diabetes or hypertension
* Regular resident of the Philadelphia metro area without plans to leave in the next 6 months

Exclusion Criteria:

* Does not meet all of the inclusion criteria
* Unable to provide consent
* Non-English speaker
* Cognitive impairment, per principal investigators' discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Richterman, MD, MPH, Principal Investigator — University of Pennsylvania; Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,132 individuals were contacted via the electronic health portal. 242 completed the interest form, and of those 142 were excluded due to ineligibility, not interested, unable to contact or unable to schedule. 100 were enrolled and randomized.
Period: Overall Study
Arm/Group | Control | Cash Transfer
Started | 50 | 50
Completed | 44 | 49
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Cash Transfer | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (9.9) | 48.5 (11.5) | 46.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 50 | 47 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 45 | 90
  White | 2 | 2 | 4
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Sexual Orientation [Count of Participants; unit: Participants]
  Straight/Heterosexual | 42 | 47 | 89
  LGBTQ+ | 7 | 2 | 9
  Prefer not to say | 1 | 1 | 2
BMI [Count of Participants; unit: Participants]
  Obesity | 44 | 39 | 83
  Overweight | 5 | 10 | 15
  Healthy | 1 | 1 | 2
Household Income [Count of Participants; unit: Participants]
  Less than $10,000 | 14 | 10 | 24
  $10,000 to $14,999 | 11 | 7 | 18
  $15,000 to $24,999 | 9 | 9 | 18
  $25,000 to $34,999 | 6 | 11 | 17
  $35,000 to $49,999 | 5 | 9 | 14
  $50,000 to $74,999 | 3 | 3 | 6
  $75,000 to $99,999 | 2 | 1 | 3
Income at the Federal Poverty Level [Count of Participants; unit: Participants] — Calculated using the 2022 federal poverty levels, based on self-reported household size.
  Participants
    <50% of federal poverty level | 16 | 9 | 25
    50-75% of federal poverty level | 9 | 7 | 16
    75-100% of federal poverty level | 8 | 11 | 19
    100-133% of federal poverty level | 5 | 9 | 14
    133%+ of federal poverty level | 12 | 14 | 26
On government assistance [Count of Participants; unit: Participants]
  Yes | 36 | 35 | 71
  No | 14 | 15 | 29
Work and School [Count of Participants; unit: Participants]
  No School or Work | 27 | 23 | 50
  Work | 22 | 24 | 46
  School and Work | 1 | 3 | 4
Main income source [Count of Participants; unit: Participants]
  A Job | 23 | 27 | 50
  Disability or Social Security | 8 | 14 | 22
  Family or friends | 9 | 2 | 11
  SNAP (Food Stamps) | 6 | 4 | 10
  Unemployment | 0 | 2 | 2
  TANF (Cash Assistance/Welfare) | 2 | 0 | 2
  Veteran Benefits | 1 | 1 | 2
  Hustling (e.g., petty theft) | 1 | 0 | 1
For those with ANY income from a job over the past 3 months (n=52), number of hours worked [Mean (Standard Deviation); unit: Hours] — This question was asked of the 52 people who reported having ANY income from a job over the past 3 months. This is in contrast to the 50 people for whom a job was the MAIN source of income over the past 3 months, and the 50 people who reported CURRENTLY having a job. Population: For those who reported source of income as "a job" (n=52)
  Hours
    number analyzed (Participants) | 25 | 27 | 52
    (all) | 30.8 (17.8) | 37.3 (13.3) | 34.1 (15.6)
Type of job [Count of Participants; unit: Participants] — This question was asked of the 52 people who reported having ANY income from a job over the past 3 months. This is in contrast to the 50 people for whom a job was the MAIN source of income over the past 3 months, and the 50 people who reported CURRENTLY having a job. Population: For those who selected "a job" for source of income (n=52)
  Participants
    number analyzed (Participants) | 25 | 27 | 52
    For Profit Org/Company | 11 | 13 | 24
    Other | 7 | 8 | 15
    Government (Local, State, Federal) | 3 | 4 | 7
    Non-Profit Org | 3 | 2 | 5
    Owner non-incorporated business | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  Less than HS | 4 | 2 | 6
  Completed HS/GED | 21 | 15 | 36
  Some College | 11 | 15 | 26
  Associates/Bachelors+ | 14 | 18 | 32
Marital status [Count of Participants; unit: Participants]
  Single | 29 | 29 | 58
  Married/Partnered | 13 | 10 | 23
  Widow/Divorced/Separated | 8 | 11 | 19
Number of people in household [Mean (Standard Deviation); unit: Number of people in household] | 2.8 (1.7) | 3.1 (2.3) | 3.0 (2.0)
Kids in household [Count of Participants; unit: Participants]
  Yes | 27 | 24 | 51
  No | 23 | 26 | 49
Living situation [Count of Participants; unit: Participants]
  Rent | 32 | 24 | 56
  Own | 8 | 15 | 23
  Elsewhere | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Food Security Category
Description: Change from baseline in food security in the last 30 days as measured by the US Department of Agriculture food security scale. Outcome is 3 ordered categories: high or marginal food security, low food security, very low food security.
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Population: 100 enrolled participants at baseline and 93 participants at 3-month follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Cash Transfer Baseline; Cash Transfer Follow-up: Participants will receive $125 every 2 weeks for 8 payments via ClinCard, for a total of $1000.
  Cash Transfer: Participants will receive $125 every 2 weeks for 8 payments via ClinCard, for a total of $1000.
- Control Baseline; Control Follow-up: No intervention
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
Participants
  High or marginal | 27 | 19 | 16 | 23
  Low | 6 | 15 | 18 | 7
  Very low | 17 | 14 | 14 | 13
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — All panel-data marginal models use robust standard errors. Categorical outcomes were assessed with ordered logistic models and continuous outcomes were assessed with GEE population-averaged models, except Medication Expenditures which used Poisson models to account for count data. Some outcomes are missing additional data (not >10%); Odds Ratio (OR) = 3.24, 95% CI 2-sided [0.84 to 12.55]

2. Primary Outcome: Change in Utility Security Category
Description: Change from baseline in utility security in the last 3 months as measured by the Home Energy Insecurity scale. Outcome is 5 ordered categories: thriving, capable, stable, vulnerable, in-crisis.
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 48 | 50 | 43
Participants
  In-crisis | 19 | 15 | 17 | 14
  Vulnerable | 11 | 11 | 10 | 7
  Stable | 9 | 9 | 11 | 7
  Capable | 8 | 5 | 8 | 5
  Thriving | 3 | 8 | 4 | 10
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.24 to 2.64]

3. Primary Outcome: Change in Financial Well-being Scale
Description: Change from baseline in current financial well-being as measured by the Consumer Financial Protection Bureau Financial Well-Being 0-100 scale (higher scores are correlated to more well-being).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
scores on a scale | 44 (12) | 44 (10) | 47 (11) | 46 (13)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.52, 95% CI 2-sided [-3.78 to 4.82]

4. Primary Outcome: Change in Perceived Stress Scale
Description: Change from baseline in perceived stress in the last 30 days as measured by the Perceived Stress Scale (short form; 0-16, higher scores are correlated to more stress).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 7.2 (3.2) | 7.1 (3.1) | 7.4 (3.3) | 7.0 (3.4)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — All panel-data marginal models use robust standard errors. The binary outcome, Future Preference: Behavioral task was assessed with a logistic model and continuous outcomes were assessed with GEE population-averaged models, except All Health Care Expenditures which used Poisson models to account for count data. Some outcomes are missing additional data (not >10%); Mean Difference (Net) = 0.20, 95% CI 2-sided [-1.01 to 1.40]

5. Primary Outcome: Change in State Anxiety Scale
Description: Change from baseline in current anxiety as measured by the State Trait Anxiety Inventory subscale. The range is from 20-80 with lower scores meaning less anxiety.
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 38 (14) | 35 (12) | 40 (13) | 41 (13)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = -2.71, 95% CI 2-sided [-7.43 to 2.00]

6. Primary Outcome: Change in Mental Bandwidth
Description: Change from baseline in number of lapses in the Psychomotor Vigilance Task (more lapses indicate less mental bandwidth).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: Change in Lapses
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
Change in Lapses | 9.0 (12) | 8.8 (13) | 11.1 (16) | 12.0 (13)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.65, 95% CI 2-sided [-5.45 to 4.16]

7. Primary Outcome: Change in Health Care Expenditures on Medications
Description: Change from baseline in number of dollars spent out-of-pocket on medications in the past 30 days.
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
Dollars | 12 (21) | 23 (45) | 10 (15) | 18 (48)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; IRR = 1.12, 95% CI 2-sided [0.46 to 2.74]

8. Primary Outcome: Change in Adherence to Medication Refills Scale
Description: Change from baseline in current adherence to refilling medications as measured by that subscale of the Adherence to Refills and Medications Scale (ARMS; 4-16, higher scores indicate lower adherence).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 6.9 (1.4) | 6.6 (1.1) | 6.5 (1.1) | 6.9 (1.3)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.75, 95% CI 2-sided [-1.29 to -0.21]

9. Secondary Outcome: Change in Number of Emergency Department Visits
Description: We had initially hoped to descriptively summarize these outcomes as part of this pilot study, but the staff member leading our analyses departed during the course of this study and we no longer had someone with the skills and bandwidth to pull, merge, and analyze these data from the electronic health record. For that reason, the data were never collected in this sample and so we have not reported these outcomes
Time Frame: Once all study appointments are completed, ED visit data will be collected through the Data Analytics Center for the 3-month period before baseline, and the 3-month period after baseline.
Reporting Status: Not Posted

10. Secondary Outcome: Change in Number of Health Care Visits (Non-emergency Department)
Description: as for outcome 9
Time Frame: Once all study appointments are completed, number of health care visits(non-ED) data will be collected through the Data Analytics Center for the 3-month period before baseline, and the 3-month period after baseline.
Reporting Status: Not Posted

11. Secondary Outcome: Change in Cigarette Dependence Scale
Description: Change from baseline in current cigarette dependence as measured by the Cigarette Dependence Scale (short version; 5-25, higher scores indicate more dependence).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 14 (4) | 15 (4) | 14 (4) | 14 (4)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.57, 95% CI 2-sided [-1.90 to 3.03]

12. Secondary Outcome: Change in Alcohol Use Scale
Description: Change from baseline in current alcohol use as measured by the Alcohol Use Disorders Identification Test (0-12, higher scores indicate more use).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 1.5 (1.6) | 1.6 (1.5) | 1.5 (1.8) | 1.5 (1.7)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.32 to 0.58]

13. Secondary Outcome: Change in All Health Care Expenditures
Description: Change from baseline in sum of dollars spent out-of-pocket on medications, office visits, and emergency room visits in the past 30 days.
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
dollars | 19 (31) | 35 (73) | 12 (17) | 35 (87)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; IRR = 0.62, 95% CI 2-sided [0.23 to 1.63]

14. Secondary Outcome: Change in Time Preference (Patience)
Description: Change from baseline on current patience which is a single item in the Preference Survey Module (0 "completely unwilling" to 10 "completely willing" to give up present benefits for future benefits, higher scores indicate future preference).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 6.8 (3.5) | 8 (2.7) | 6.5 (3.5) | 6.7 (3.2)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = 1.05, 95% CI 2-sided [-0.54 to 2.64]

15. Secondary Outcome: Change in Time Preference (Behavioral Task)
Description: Change from baseline on current snack choice (binary: chose a more or a less healthy snack, choosing a healthy snack indicates future preference).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
Participants
  Selected Fruit | 40 | 27 | 33 | 20
  Selected Snack | 7 | 15 | 12 | 21
  No Selection | 3 | 7 | 5 | 3
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.19 to 5.49]

16. Secondary Outcome: Change in Psychological Distress Scale
Description: Change from baseline in psychological distress in the past 30 days as measured by the Kessler Psychological Distress Scale (K6+, 6-30, higher scores indicate more distress).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 13 (6) | 12 (5) | 13 (6) | 14 (5)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = -1.10, 95% CI 2-sided [-2.64 to 0.43]

17. Secondary Outcome: Change in Number of Healthy Days
Description: Change from baseline in self-reported number of healthy days in the past 30 as measured by the CDC Health-Related Quality of Life Scale (0-30 days).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
days | 12 (11) | 15 (11) | 14 (11) | 15 (11)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = 2.72, 95% CI 2-sided [-1.35 to 6.80]

18. Secondary Outcome: Change in Adherence to Taking Medications Scale
Description: Change from baseline in current adherence to taking medications as measured by that subscale of the Adherence to Refills and Medications Scale (ARMS; 8-32, higher scores indicate lower adherence).
Time Frame: Assessed at 1-hour appointment at baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
Number analyzed (Participants) | 50 | 49 | 50 | 44
score on a scale | 11 (3) | 10 (2) | 11 (3) | 11 (3)
Statistical Analysis 1: Comparison: Cash Transfer Baseline vs Cash Transfer Follow-up vs Control Baseline vs Control Follow-up; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.69, 95% CI 2-sided [-1.74 to 0.36]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Cash Transfer Baseline | Cash Transfer Follow-up | Control Baseline | Control Follow-up
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/50 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/50 | 0/44
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/50 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05838027/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT05838027/SAP_001.pdf